CLINICAL TRIAL: NCT03132142
Title: Temporal Profile of the Nociceptive Desensitization Induced by 8% Topical Capsaicin and the Functional Independence of Transient Receptor Potential Ankyrin 1 (TPRA1)- and Vanilloid 1 (TRPV1)-Expressing Nociceptive Afferents
Brief Title: Desensitization of Nociceptive Afferents by Application of Topical Capsaicin, Trans-cinnamaldehyde and L-menthol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Hjalte Holm Andersen, MSc. Med., Phd. Stud., Aalborg University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: N-20170018
Record Dates: First submitted 2017-04-25; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Pain; Pruritus; Neuropathic Pain; Dermatology/Skin - Other
MeSH Terms: conditions — Pain; Pruritus; Neuralgia | interventions — Capsaicin; cinnamaldehyde; Menthol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Capsaicin (Experimental): Capsacin (8%) patches applied topically 4 times for 1 hour to a 4x4 cm predefined area on the skin of the volar forearms.
  Interventions: Drug: Capsaicin
- Trans-cinnamaldehyde (Experimental): Trans-cinnamaldehyde (10%, dissolved in 90% ethanol) applied topically 4 times for 1 hour to a 4x4 cm predefined area on the skin of the volar forearms on a cotton ball placed in a plastic chamber to limit evaporation.
  Interventions: Drug: Trans-cinnamaldehyde
- L-menthol (Experimental): L-menthol (40%, dissolved in 96% ethanol) applied topically 4 times for 1 hour to a 4x4 cm predefined area on the skin of the volar forearms on a cotton ball placed in a plastic chamber to limit evaporation.
  Interventions: Drug: L-Menthol
- Vehicle patch (Placebo Comparator): Inert vehicle patches applied topically 4 times for 1 hour to a 4x4 cm predefined area on the skin of the volar forearms.
  Interventions: Drug: Vehicle patch

INTERVENTIONS:
Drug: Capsaicin — 4x4 cm patch of 8% topical capsaicin applied to the skin of the volar forearm for 1 hour 4 times on 4 consecutive days
  Arms: Capsaicin
Drug: Trans-cinnamaldehyde — 1mL of 10% trans-cinnamaldehyde applied to the skin of the volar forearm for 1 hour 4 times on 4 consecutive days
  Arms: Trans-cinnamaldehyde
Drug: L-Menthol — 1mL of 40% L-menthol applied to the skin of the volar forearm for 1 hour 4 times on 4 consecutive days
  Arms: L-menthol
Drug: Vehicle patch — Inert vehicle patch applied to the skin of the volar forearm for 1 hour 4 times on 4 consecutive days
  Arms: Vehicle patch

SUMMARY:
The purpose of this study is to investigate the potential desensitising effects of repeated applications of capsaicin, trans-cinnamaldehyde and L-menthol on thermal, mechanical and chemical sensory stimulations.

DETAILED DESCRIPTION:
Capsaicin, the compound responsible for the pungency of chili peppers, can induce desensitization to nociceptive (1) and pruriceptive (2) stimuli when topically applied. The purpose of this study is to determine whether repeated topical applications of trans-cinnamaldehyde and L-menthol result in decreased responses to various nociceptive and non-nociceptive thermal and mechanical stimuli and to compare potential alterations with those caused by repeated topical application of capsaicin. Furthermore, this study investigates the temporal profile of said alterations.

Capsaicin 8% patches, trans-cinnamaldehyde 10%, L-menthol 40% and inert vehicle patches will each be applied to 4 4x4 cm predefined areas on the skin of the volar forearms for 1 hour 4 times on 4 consecutive days. Before each application and the day after the last application, cold detection threshold (CDT), warmth detection threshold (WDT), cold pain threshold (CPT) and heat pain threshold (HPT) will be assessed using a Medoc Pathway (Medoc, Israel) equipped with a 3x3 cm contact thermode. On the last day, mechanical detection threshold (MDT) is assessed using a series of von Frey filaments and mechanical pain threshold (MPT) and mechanical pain sensitivity (MPS) is assessed using a series of standardized pinprick stimulators (Aalborg University).

Furthermore, full-field laser perfusion imaging (FLPI) will be used to assess the degree of neurogenic inflammation in each predefined area before and after each substance application and at the last session.

1. F. Henrich et al. 2015 "Capsaicin-sensitive C- and A-fibre nociceptors control long-term potentiation-like pain amplification in humans"
2. H.H. Andersen et al. 2017 "Antipruritic effect of pretreatment with 8% topical capsaicin on histamine- and cowhage-evoked itch in healthy volunteers - a randomized placebo-blinded proof-of-concept trial"

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Speaks and understands English or Danish
* 18-60 years

Exclusion Criteria:

* Pregnancy or lactation
* Drug addiction
* Previous or current dermatological, neurological, musculoskeletal or mental illnesses
* Lack of ability to cooperate
* Current use of medications that may affect the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Cold Pain Threshold (CPT) | Assessed at 5 visits on 5 consecutive days
  The pain threshold for cold stimulation assessed using a Medoc Pathway (Medoc, Israel) equipped with a 3x3 cm thermode. CPT is defined as the temperature at which cold induces pain and is expressed in °C.
Heat Pain Threshold (HPT) | Assessed at 5 visits on 5 consecutive days
  The pain threshold for heat stimulation

SECONDARY OUTCOMES:
Neurogenic Inflammation Intensity | Assessed before and after application of substances at 5 visits on 5 consecutive days
  The average intensity of the neurogenic inflammation as assessed by full-field laser perfusion imaging (FLPI) (expressed in arbitrary units)
Neurogenic Inflammation Area | Assessed before and after application of substances at 5 visits on 5 consecutive days
  The area of the neurogenic inflammation as assessed by full-field laser perfusion imaging (FLPI) (expressed in arbitrary units)
Pain During Application of Capsaicin | Assessed every 5 minutes during the 60 minute application of capsaicin at 4 visits on 4 consecutive days
  Pain during the 60 minute application of topical capsaicin as rated on a visual analog scale (VAS) (0-10)
Pain During Application of Trans-cinnamaldehyde | Assessed every 5 minutes during the 60 minute application of trans-cinnamaldehyde at 4 visits on 4 consecutive days
  Pain during the 60 minute application of trans-cinnamaldehyde as rated on a visual analog scale (VAS) (0-10)
Pain During Application of L-menthol | Assessed every 5 minutes during the 60 minute application of L-menthol at 4 visits on 4 consecutive days
  Pain during the 60 minute application of L-menthol as rated on a visual analog scale (VAS) (0-10)
Pain During Application of Inert Patch (Control) | Assessed every 5 minutes during the 60 minute application of the inert patch (control) at 4 visits on 4 consecutive days
  Pain during the 60 minute application of the inert patch (control) as rated on a visual analog scale (VAS) (0-10)
Cold Detection Threshold (CDT) | Assessed at 5 visits on 5 consecutive days
  The detection threshold for cold stimulation assessed using a Medoc Pathway (Medoc, Israel) equipped with a 3x3 cm thermode. CDT is defined as the temperature at which cold can be detected and is expressed in °C.
Warmth Detection Threshold (WDT) | Assessed at 5 visits on 5 consecutive days
  The detection threshold for warmth stimulation assessed using a Medoc Pathway (Medoc, Israel) equipped with a 3x3 cm thermode. WDT is defined as the temperature at which warmth can be detected and is expressed in °C.
Mechanical Detection Threshold (MDT) | Assessed at day 5 (final visit)
  The detection threshold for mechanical stimulation is defined as the smallest force that can be felt and is assessed using a series of standardized von Frey filaments and using the "method of limits" employing a series of stimulations with ascending and descending force expressed in mN.
Mechanical Pain Threshold (MPT) | Assessed at day 5 (final visit)
  The pain threshold for mechanical stimulation is defined as the smallest force that induces pain and is assessed using a series of standardized pinprick stimulators (Aalborg University) and using the "method of limits" employing a series of stimulations with ascending and descending forces expressed in mN.
Mechanical Pain Sensitivity (MPS) | Assessed at day 5 (final visit)
  The sensitivity to mechanically induced pain induced by a series of 7 standardized pinprick stimulators (Aalborg University) as rated on a visual analog scale (VAS) ranging from 0-10 with 0 representing no pain and 10 representing the worst pain imaginable.
Vibration Detection Threshold | Assessed at day 5 (final visit)
  The detection threshold for vibrational stimulation assessed using a Vibrameter (Somedic, Sweden).

CONTACTS AND LOCATIONS:
Locations (1):
- SMI, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No